CLINICAL TRIAL: NCT02571322
Title: The Effect of Whole Body Vibration Training on Body Composition, Physical Fitness, and Quality of Life
Brief Title: Whole Body Vibration Training on Body Composition
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding; logistics of conducting study were very complex.
Sponsor: University of Miami (Other)
Collaborators: HyperVibe Pty Ltd (Industry)
Responsible Party: Principal Investigator, John E. Lewis, Principal Investigator, University of Miami
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 20150524
Record Dates: First submitted 2015-09-28; First posted 2015-10-08 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Body Composition, Beneficial; Physical Fitness
MeSH Terms: conditions — Glucocorticoid Receptor Deficiency | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Whole Body Vibration training (Experimental): Use of the HyperVibe Whole Body Vibration training device for 12 weeks 3 times per week crossover to aerobic exercise
  Interventions: Device: HyperVibe Whole Body Vibration training device
- Aerobic Exercise (Placebo Comparator): Aerobic exercise training for 12 weeks 3 times per week crossover to use of the HyperVibe Whole Body Vibration training device
  Interventions: Other: Aerobic Exercise

INTERVENTIONS:
Device: HyperVibe Whole Body Vibration training device — Standing on the HyperVibe platform during WBV training will cause repetitive upward movements of platform to be felt by participant.Thus the participant will feel a whole body vibration, as the name of training implies. Each session will last approximately fifteen minutes.
  Arms: Whole Body Vibration training
Other: Aerobic Exercise — Aerobic exercise session will last approximately thirty minutes. Starting training intensity will be specific to each participant based on his/her baseline fitness level.
  Arms: Aerobic Exercise

SUMMARY:
The purpose of the study is to determine the effect of whole-body vibration (WBV) on body composition, physical fitness, and quality of life.

DETAILED DESCRIPTION:
The purpose of the study is to determine the effect of whole-body vibration (WBV) on body composition, physical fitness, and quality of life.Twenty healthy adult males and females (ages 18-65) with no contraindications for exercise training will be recruited to participate in the study. Subjects will participate in a randomized, crossover trial for 24 weeks. Subjects will be assigned to either: (1) WBV for the first 12 weeks and then aerobic exercise training for the second 12 weeks 3 times per week (n=10) or (2) aerobic exercise training for the first 12 weeks and then WBV for the second 12 weeks 3 times per week (n=10). Subjects will be assessed at baseline and at 12 and 24 weeks on aerobic capacity (estimated VO2max), upper and lower body strength (1-repetition maximum on bench press and leg press, respectively), compartmental and total body fat mass, fat free mass, and bone mineral density (using dual energy x-ray absorptiometry (DEXA)), body mass index (height relative to weight), weight, skin fold and body part circumferences, resting blood pressure and pulse, and subjective health-related quality of life (SF-36). Participants will be trained and assessed at the University of Miami Miller School of Medicine UHealth Fitness and Wellness Center, in UHealth Champions Executive Medicine, and in the Department of Psychiatry and Behavioral Sciences.

No substantial psychological, medical, or social risks exist to the participants. Although all measures to protect confidentiality will be put in place, the possibility exists that electronic data could be jeopardized. In the remote case that such event occurs, it will be immediately reported to the Institutional Review Board (IRB).

Exercise has been shown to be safe among every population, including those with chronic diseases and/or other complications. A DEXA scan is the equivalent of about 4 extra days' worth of naturally-occurring radiation.

The use of the HyperVibe WBV training device should be harmless without any known negative effects, as WBV is even lower risk than aerobic exercise, as the participant simply stands on the platform without moving while being exposed to full-body vibration. The system is completely non-invasive, and no serious, untoward side effects have been reported to the manufacturer (HyperVibe) of this system. All study personnel will follow instructions for operating the system. Participants will incur no additional appreciable psychological or social risks by participating in this study.

The results obtained in this study may demonstrate a way to increase exercise efficiency through the use of WBV in helping overweight/obese participants to lose weight, gain muscular weight, and improve physical fitness levels. By participating in the study, subjects may improve their overall health status in a unique approach to exercise training. The minimal risk of participating in this study is reasonable because the potential information gained can be worthwhile for helping people to lose weight, which is significant, given the inordinate prevalence of overweight/obesity and its co morbid chronic diseases in the United States today.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ages 18 to 65 years old
2. Interest in participating in a study to investigate the effects of a novel exercise training style
3. Willing to follow recommendations for participating in the study
4. Able to provide informed consent to participate in the study

Exclusion Criteria:

1. Women who are pregnant or attempting pregnancy during the next 24 weeks
2. Anyone with a cardiovascular, orthopedic, or other physical condition that would be contraindicated for an exercise training program
3. Any condition where WBV is contraindicated, e.g., seizure disorder
4. Currently enrolled in another exercise intervention research study
5. Currently undergoing internal defibrillation, like with an implantable heart device
6. Erratic, accelerated, or mechanically controlled irregular heart rhythms
7. Atrial fibrillation/flutter
8. Atrioventricular block
9. Recently had dyes introduced into the bloodstream, such as methylene blue, indocyanine green, indigo carmine, and fluorescein
10. Any implanted electronic device

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01-19 (Actual); Primary Completion 2017-01-12 (Actual); Study Completion 2017-01-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in body composition | Baseline,12 weeks and 24 weeks
  Body composition will be evaluated by DEXA scan which measure fat free mass , total body and compartmental fat mass
Change from baseline in aerobic capacity | Baseline,12 weeks and 24 weeks
  Aerobic capacity and strength will be assessed by Graded Exercise Test
Change from baseline in body strength | Baseline,12 weeks and 24 weeks
  Overall upper and lower body strength will be assessed by one-repetition maximum strength tests
Change from baseline in bone mineral density | Baseline,12 weeks and 24 weeks
  Bone mineral density will be assessed by DEXA scan

SECONDARY OUTCOMES:
Change from baseline in physical activity | Baseline,12 weeks and 24 weeks
  Physical activity will be assessed with International Physical Activity Questionnaire (IPAQ). The IPAQ items are structured to provide individual domain specific scores for walking, moderate-intensity, and vigorous activity within the domains of work, transportation, domestic chores and gardening, and leisure-time. The tool asks about the time spent doing a specific physical activity in the last 7 days. For total scores, the duration (in minutes) and frequency for all types of activities in all domains are summed, while specific domain scores are calculated by the summation of the walking, moderate-intensity and vigorous-intensity activities within the specific domain. For activity-specific scores, the scores for the specific type of activity across domains are added. To measure the volume of activity, each type of activity is weighted by its energy requirement defined as the metabolic equivalent of task-minute (MET-min).
Change from baseline in quality of life | Baseline,12 weeks and 24 weeks
  The SF-36 (v2) Health Survey provides psychometrically-based physical and mental health summary measures and a preference-based health utility index. It is a generic measure that does not target a specific age, disease, or treatment group.
Change from baseline in systolic blood pressure | Baseline,12 weeks and 24 weeks
  Systolic blood pressure will be measured to the nearest even digit by use of the Microlife Deluxe upper arm blood pressure monitor. Three readings will be made with the subjects seated after they have rested for five minutes. The average of the three readings will be used in the analysis
Change from baseline in diastolic blood pressure | Baseline,12 weeks and 24 weeks
  Diastolic blood pressure will be measured to the nearest even digit by use of the Microlife Deluxe upper arm blood pressure monitor. Three readings will be made with the subjects seated after they have rested for five minutes. The average of the three readings will be used in the analysis

CONTACTS AND LOCATIONS:
Overall Officials: John E Lewis, Ph.D., Principal Investigator — University of Miami
Locations (1):
- University of Miami Miller School of Medicine, Clinical Research Building, Department of Psychiatry & Behavioral Sciences, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adcox, S (2002, September 21). New state law seeks to cut down obesity. Ithaca Journal.
- [Background] Baumgartner RN, Roche AF, Guo S, Lohman T, Boileau RA, Slaughter MH. Adipose tissue distribution: the stability of principal components by sex, ethnicity and maturation stage. Hum Biol. 1986 Oct;58(5):719-35. No abstract available. PMID 3804294
- [Background] Bautmans I, Van Hees E, Lemper JC, Mets T. The feasibility of Whole Body Vibration in institutionalised elderly persons and its influence on muscle performance, balance and mobility: a randomised controlled trial [ISRCTN62535013]. BMC Geriatr. 2005 Dec 22;5:17. doi: 10.1186/1471-2318-5-17. PMID 16372905
- [Background] Bosco C, Colli R, Introini E, Cardinale M, Tsarpela O, Madella A, Tihanyi J, Viru A. Adaptive responses of human skeletal muscle to vibration exposure. Clin Physiol. 1999 Mar;19(2):183-7. doi: 10.1046/j.1365-2281.1999.00155.x. PMID 10200901
- [Background] Bruyere O, Wuidart MA, Di Palma E, Gourlay M, Ethgen O, Richy F, Reginster JY. Controlled whole body vibration to decrease fall risk and improve health-related quality of life of nursing home residents. Arch Phys Med Rehabil. 2005 Feb;86(2):303-7. doi: 10.1016/j.apmr.2004.05.019. PMID 15706558
- [Background] Centers for Disease Control and Prevention. (2014). National diabetes statistics report Atlanta, GA: U.S. Department of Health and Human Services, Centers for Disease Control and Prevention.
- [Background] Cheung WH, Mok HW, Qin L, Sze PC, Lee KM, Leung KS. High-frequency whole-body vibration improves balancing ability in elderly women. Arch Phys Med Rehabil. 2007 Jul;88(7):852-7. doi: 10.1016/j.apmr.2007.03.028. PMID 17601464
- [Background] Church TS, Kampert JB, Gibbons LW, Barlow CE, Blair SN. Usefulness of cardiorespiratory fitness as a predictor of all-cause and cardiovascular disease mortality in men with systemic hypertension. Am J Cardiol. 2001 Sep 15;88(6):651-6. doi: 10.1016/s0002-9149(01)01808-2. PMID 11564389
- [Background] Cochrane DJ, Stannard SR, Sargeant AJ, Rittweger J. The rate of muscle temperature increase during acute whole-body vibration exercise. Eur J Appl Physiol. 2008 Jul;103(4):441-8. doi: 10.1007/s00421-008-0736-4. PMID 18392845
- [Background] Colditz GA. Economic costs of obesity and inactivity. Med Sci Sports Exerc. 1999 Nov;31(11 Suppl):S663-7. doi: 10.1097/00005768-199911001-00026. PMID 10593542
- [Background] Cormie P, Deane RS, Triplett NT, McBride JM. Acute effects of whole-body vibration on muscle activity, strength, and power. J Strength Cond Res. 2006 May;20(2):257-61. doi: 10.1519/R-17835.1. PMID 16686550
- [Background] Da Silva ME, Fernandez JM, Castillo E, Nunez VM, Vaamonde DM, Poblador MS, Lancho JL. Influence of vibration training on energy expenditure in active men. J Strength Cond Res. 2007 May;21(2):470-5. doi: 10.1519/R-19025.1. PMID 17530948
- [Background] Dastmenash, S., van den Tillaar, R., Jacobs, P., Shafiee, G., & Shojaedin, S. (2010). The effect of whole body vibration, PNF training or a combination of both on hamstrings range of motion. World Applied Sciences Journal, 11, 744-751
- [Background] Di Pietro L, Dziura J, Blair SN. Estimated change in physical activity level (PAL) and prediction of 5-year weight change in men: the Aerobics Center Longitudinal Study. Int J Obes Relat Metab Disord. 2004 Dec;28(12):1541-7. doi: 10.1038/sj.ijo.0802821. PMID 15543159
- [Background] Ditschuneit HH, Flechtner-Mors M. Value of structured meals for weight management: risk factors and long-term weight maintenance. Obes Res. 2001 Nov;9 Suppl 4:284S-289S. doi: 10.1038/oby.2001.132. PMID 11707555
- [Background] Flegal KM, Carroll MD, Kit BK, Ogden CL. Prevalence of obesity and trends in the distribution of body mass index among US adults, 1999-2010. JAMA. 2012 Feb 1;307(5):491-7. doi: 10.1001/jama.2012.39. Epub 2012 Jan 17. PMID 22253363
- [Background] Flegal KM, Carroll MD, Ogden CL, Johnson CL. Prevalence and trends in obesity among US adults, 1999-2000. JAMA. 2002 Oct 9;288(14):1723-7. doi: 10.1001/jama.288.14.1723. PMID 12365955
- [Background] Guo Y, Franks PW, Brookshire T, Antonio Tataranni P. The intra- and inter-instrument reliability of DXA based on ex vivo soft tissue measurements. Obes Res. 2004 Dec;12(12):1925-9. doi: 10.1038/oby.2004.241. PMID 15687392
- [Background] Haapanen N, Miilunpalo S, Pasanen M, Oja P, Vuori I. Association between leisure time physical activity and 10-year body mass change among working-aged men and women. Int J Obes Relat Metab Disord. 1997 Apr;21(4):288-96. doi: 10.1038/sj.ijo.0800403. PMID 9130026
- [Background] Helmrich SP, Ragland DR, Leung RW, Paffenbarger RS Jr. Physical activity and reduced occurrence of non-insulin-dependent diabetes mellitus. N Engl J Med. 1991 Jul 18;325(3):147-52. doi: 10.1056/NEJM199107183250302. PMID 2052059
- [Background] Hill JO, Wyatt HR, Reed GW, Peters JC. Obesity and the environment: where do we go from here? Science. 2003 Feb 7;299(5608):853-5. doi: 10.1126/science.1079857. PMID 12574618
- [Background] Klem ML, Wing RR, McGuire MT, Seagle HM, Hill JO. A descriptive study of individuals successful at long-term maintenance of substantial weight loss. Am J Clin Nutr. 1997 Aug;66(2):239-46. doi: 10.1093/ajcn/66.2.239. PMID 9250100
- [Background] Leermakers EA, Perri MG, Shigaki CL, Fuller PR. Effects of exercise-focused versus weight-focused maintenance programs on the management of obesity. Addict Behav. 1999 Mar-Apr;24(2):219-27. doi: 10.1016/s0306-4603(98)00090-2. PMID 10336103
- [Background] Lewis, J. & Schneiderman, N. (2006). Nutrition, physical activity, weight management, and health. Revista Colombiana de Psiquiatría, 35, 157S-175S
- [Background] Ogden CL, Carroll MD, Kit BK, Flegal KM. Prevalence of obesity in the United States, 2009-2010. NCHS Data Brief. 2012 Jan;(82):1-8. PMID 22617494
- [Background] Pasman WJ, Saris WH, Muls E, Vansant G, Westerterp-Plantenga MS. Effect of exercise training on long-term weight maintenance in weight-reduced men. Metabolism. 1999 Jan;48(1):15-21. doi: 10.1016/s0026-0495(99)90004-5. PMID 9920139
- [Background] Pasman WJ, Saris WH, Westerterp-Plantenga MS. Predictors of weight maintenance. Obes Res. 1999 Jan;7(1):43-50. doi: 10.1002/j.1550-8528.1999.tb00389.x. PMID 10023729
- [Background] Pi-Sunyer, F., Becker, D., Bouchard, C., & Carlton, R. (1998). NHLBI obesity education initiative expert panel on the identification, evaluation, and treatment of overweight and obesity in adults. Obesity Research, 6, 51S-209S.
- [Background] Powers Hannley P. Move more, eat less: it's time for Americans to get serious about exercise. Am J Med. 2014 Aug;127(8):681-4. doi: 10.1016/j.amjmed.2014.05.026. Epub 2014 Jun 6. No abstract available. PMID 24909130
- [Background] Ronnestad BR. Acute effects of various whole body vibration frequencies on 1RM in trained and untrained subjects. J Strength Cond Res. 2009 Oct;23(7):2068-72. doi: 10.1519/JSC.0b013e3181b8652d. PMID 19855332
- [Background] Ronnestad BR. Acute effects of various whole-body vibration frequencies on lower-body power in trained and untrained subjects. J Strength Cond Res. 2009 Jul;23(4):1309-15. doi: 10.1519/JSC.0b013e318199d720. PMID 19568035
- [Background] Rubin C, Recker R, Cullen D, Ryaby J, McCabe J, McLeod K. Prevention of postmenopausal bone loss by a low-magnitude, high-frequency mechanical stimuli: a clinical trial assessing compliance, efficacy, and safety. J Bone Miner Res. 2004 Mar;19(3):343-51. doi: 10.1359/JBMR.0301251. Epub 2003 Dec 22. PMID 15040821
- [Background] Schmitz KH, Jacobs DR Jr, Leon AS, Schreiner PJ, Sternfeld B. Physical activity and body weight: associations over ten years in the CARDIA study. Coronary Artery Risk Development in Young Adults. Int J Obes Relat Metab Disord. 2000 Nov;24(11):1475-87. doi: 10.1038/sj.ijo.0801415. PMID 11126345
- [Background] Sturm R. The effects of obesity, smoking, and drinking on medical problems and costs. Health Aff (Millwood). 2002 Mar-Apr;21(2):245-53. doi: 10.1377/hlthaff.21.2.245. PMID 11900166
- [Background] United States Department of Health and Human Services. (1996). Physical Activity and Health: A Report of the Surgeon General (Rep. No. 017-023-00196-5). Atlanta, GA: United States Department of Health and Human Services, Centers for Disease Control and Prevention, National Center for Chronic Disease Prevention and Health Promotion.
- [Background] United States Department of Health and Human Services. (2000). Healthy people 2010: Understanding and improving health Washington, DC: United States Government Printing Office.
- [Background] United States Department of Health and Human Services. (2010). Healthy people 2020 Washington, DC: United States Government Printing Office.
- [Background] Office of the Surgeon General (US); Office of Disease Prevention and Health Promotion (US); Centers for Disease Control and Prevention (US); National Institutes of Health (US). The Surgeon General's Call To Action To Prevent and Decrease Overweight and Obesity. Rockville (MD): Office of the Surgeon General (US); 2001. Available from http://www.ncbi.nlm.nih.gov/books/NBK44206/ PMID 20669513
- [Background] Visscher TL, Seidell JC. The public health impact of obesity. Annu Rev Public Health. 2001;22:355-75. doi: 10.1146/annurev.publhealth.22.1.355. PMID 11274526
- [Background] Ware, J., Kosinski, M., & Dewey, J. (2000). How to score version two of the sf-36 health survey. Lincoln, RI: QualityMetric, Inc.
- [Background] Westerterp-Plantenga MS, Kempen KP, Saris WH. Determinants of weight maintenance in women after diet-induced weight reduction. Int J Obes Relat Metab Disord. 1998 Jan;22(1):1-6. doi: 10.1038/sj.ijo.0800536. PMID 9481593
- [Background] Wickelgren I. Obesity: how big a problem? Science. 1998 May 29;280(5368):1364-7. doi: 10.1126/science.280.5368.1364. No abstract available. PMID 9634413
- [Background] Wilcock IM, Whatman C, Harris N, Keogh JW. Vibration training: could it enhance the strength, power, or speed of athletes? J Strength Cond Res. 2009 Mar;23(2):593-603. doi: 10.1519/JSC.0b013e318196b81f. PMID 19258884
- [Background] Williamson DF, Madans J, Anda RF, Kleinman JC, Kahn HS, Byers T. Recreational physical activity and ten-year weight change in a US national cohort. Int J Obes Relat Metab Disord. 1993 May;17(5):279-86. PMID 8389337
- [Background] Obesity: preventing and managing the global epidemic. Report of a WHO consultation. World Health Organ Tech Rep Ser. 2000;894:i-xii, 1-253. PMID 11234459
- [Background] World Health Organization. (2002). Childhood nutrition and progress in implementing the international code of marketing of breast-milk substitutes (Rep. No. A55/14). Geneva.
- [Background] Zellner M. [Incontinence after radical prostatectomy and cystectomy: are combined training with mechanical devices and whole body vibration effective?]. Urologe A. 2011 Apr;50(4):433-44. doi: 10.1007/s00120-010-2478-2. German. PMID 21472620